CLINICAL TRIAL: NCT02846974
Title: Calibration and Validation of High Quality Low-Cost 3D Printed Pulse Oximeter
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other); Al Shifa Hospital, Gaza (Unknown); University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Tarek Loubani, MD, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 107952
Record Dates: First submitted 2016-07-23; First posted 2016-07-27 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Pulse Oximetry; Free and Open Source
Keywords: Pulse Oximetry; Free and Open Source

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Calibration cohort: In this cohort, approximately 30 subjects will be put through a controlled desaturation study with controlled hypoxia until they arrive at approximately SpO2 = 70%. Measurements will be taken via arterial catheterization to resolve proper values to calibrate the device
  Interventions: Device: Pulse oximeter
- Validation cohort: In this cohort, approximately 250 patients will have a single pulse oximetry reading taken using the novel device and a gold standard device to ensure accurate validation.
  Interventions: Device: Pulse oximeter

INTERVENTIONS:
Device: Pulse oximeter — A pulse oximeter will be used for calibration

SUMMARY:
Pulse oximetry is a vital tool in the rapid and non-invasive assessment of emergency patients, providing a continuous estimate of hemoglobin saturation in arterial blood. Unfortunately, the costs of these devices are prohibitive and reduce availability in smaller centres and poor countries, putting millions of patients in danger of easily treatable and preventable conditions. With current rapid prototyping technologies such as 3D printing, it is possible to create a very inexpensive pulse oximeter that meets or exceeds the gold standard. The goal of this study is to develop, validate and certify a pulse oximeter that measures hemoglobin, carboxyhemoglobin and methemoglobin. This pulse oximeter will be certified with Health Canada, and then released under the Open Hardware License (OHL), such that hospitals and ministries of health in rural and impoverished communities in Canada and internationally would have easy access to these devices.

ELIGIBILITY:
Inclusion Criteria:

- This study has 2 Phases. In Phase 1, healthy, non-smoking adult volunteers greater than 18 years of age are invited to participate. In Phase 2, all adult (>18) non-critical patients and healthy community volunteers visiting the ED at VH and UH are eligible to participate.

Exclusion Criteria:

Potential participants will be excluded based on the following criteria:

Phase 1:

* greater than 70 years of age,
* current smokers,
* previous history of cardiac disease (e.g., atrial fibrillation, myocardial infarction, congestive heart failure),
* history of moderate or severe asthma,
* history of seizures,
* history of stroke or transient ischemic attack
* pregnant women
* Patients with any active pulmonary disease such as pneumonia
* Individuals who are unwilling to participate or are less than 18 years old
* Those who are unable to consent

Phase 2

* Critical patients will be excluded from participating
* Individuals who are unwilling to participate or are less than 18 years old will be excluded
* Those who are unable to consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study has 2 Phases. In Phase 1, healthy, non-smoking adult volunteers greater than 18 years of age are invited to participate. In Phase 2, all adult (>18) non-critical patients and healthy community volunteers visiting the emergency department at Victoria Hospital and University Hospital are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulse oximetry reading | 1 hour
  Pulse oximetry readings will be taken over the span of an hour to calibrate the device
Arterial blood gas | 1 hour
  Arterial blood gases will be taken to create a proper calibration curve along with the device's readings.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Loubani, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada